CLINICAL TRIAL: NCT04128163
Title: A Twelve-month Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of QL1206 in Chinese Postmenopausal Women With Osteoporosis at High Risk of Fracture
Brief Title: Efficacy and Safety of QL1206 in the Treatment of Postmenopausal Osteoporosis With High Fracture Risk
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1206-004
Record Dates: First submitted 2019-09-25; First posted 2019-10-16 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-09

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — QL1206

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1206 (Experimental): QL1206 injection (60mg:1ml) by subcutaneous injectionevery 6 month for two times.
  Dietary Supplement: Elemental Calcium Oral, at least 500 mg Dietary Supplement: Vitamin D Oral, 1000 IU
  Interventions: Drug: QL1206
- Placebo (Placebo Comparator): placebo injection (1ml) by subcutaneous injectionevery 6 month for two times.
  Dietary Supplement: Elemental Calcium Oral, at least 500 mg Dietary Supplement: Vitamin D Oral, 1000 IU
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: QL1206 — subcutaneous injection of 60 mg（60mg:1ml）, Q6M, twice for one year.
  Dietary Supplement: Elemental Calcium Oral, at least 500 mg Dietary Supplement: Vitamin D Oral, 1000 IU
  Other Names: Recombinant anti-RANKL human monoclonal antibody injection
  Arms: QL1206
Drug: Placebos — subcutaneous injection of（1ml）, Q6M, twice for one year.
  Dietary Supplement: Elemental Calcium Oral, at least 500 mg Dietary Supplement: Vitamin D Oral, 1000 IU
  Arms: Placebo

SUMMARY:
A randomized, double-blind, two-group parallel, placebo-controlled clinical Phase III trial to compare the efficacy and safety of QL1206 and placebo in postmenopausal women with osteoporosis at high risk of fracture

DETAILED DESCRIPTION:
This is a randomized, double-blind, two-group parallel, placebo-controlled clinical Phase III trial.

The primary objective is to evaluate the effect of QL1206 treatment compared with placebo in Chinese postmenopausal women with osteoporosis at high risk of fracture.

The secondary objective is to evaluate the clinical safety, immunogenicity and pharmacokinetic (PK) characteristics of QL1206 in women with osteoporosis at high risk of postmenopausal fracture

The exploratory purpose is to evaluate the effect of ADA on the characteristics of QL1206 PK and the relationship between QL1206 exposure and pharmacodynamic endpoints, efficacy and adverse events

Subjects would sequentially enrolled according to the protocol in one of two cohorts.Subjects would receive a single 60mg of QL1206 or placebo every 6 month for1 year(twice for one, subcutaneous injection) ,meanwhile taking 500 mg of calcium and 1000IU of vitamin D daily

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing to provide written informed consent.
2. Ambulatory woman between the age of 50 and 85 years, inclusive.
3. The subject has a BMD absolute value consistent with a T-score<-2.5 and >-4.0 at either the lumbar spine or total hip
4. All subjects must have at least one of following additional the risk factors:history of fracture（after 40 years）,parental history of hip fracture, low Body mass index (BMI≤19kg/m^2), elderly (age≥65year)，current smoker
5. Postmenopausal defined as >2 years postmenopausal, which can be >2 years of spontaneous amenorrhea or >2 years post surgical bilateral oophorectomy.

Exclusion Criteria:

1. Bone/metabolic disease:a. Any metabolic bone disease, e.g., osteomalacia or osteogenesis imperfecta,which may interfere with the interpretation of the findings.

   b. Paget's disease c. Cushing's disease d. Hyperprolactinemia
2. Current hyperparathyroidism or hypoparathyroidism by medical record
3. Thyroid condition: Hyperthyroidism or hypothyroidism.
4. Rheumatoid arthritis

   -

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine from Baseline up to 12 months | Baseline and Month 12
  Bone mineral density (BMD) is the amount of bone mineral in bone tissue. BMD scan was done using dual energy x-ray absorptiometry (DXA). It is used to identify osteoporosis, determine risk for fractures, and measure response to osteoporosis treatment. The percentage change from Baseline for BMD was calcuated as the value at the indicated time point minus the Baseline value multiplied by 100 and divided by the Baseline value. The analysis was performed by Analysis of Covariance (ANCOVA) model adjusted for treatment, region and Baseline BMD for the skeletal site under consideration as a continuous covariate for assessment. Region and treatment by region interaction was included in the model. Screening visit was considered as Baseline for BMD. For participants who withdrew early, the missing BMD assessments was estimated by the Last Observation Carried Forward (LOCF), provided the assessment was taken on or after at least three month on-therapy.

SECONDARY OUTCOMES:
Percent Change in BMD at the Lumbar Spine from Baseline up to 6 months | Baseline and Month 6
  BMD is the amount of bone mineral in bone tissue. BMD scan was done using DXA. It is used to identify osteoporosis, determine risk for fractures, and measure response to osteoporosis treatment. The percentage change from Baseline for BMD was calculated as the value at the indicated time point minus the Baseline value multiplied by 100 and divided by the Baseline value
Percent change in BMD at the total hip, femoral neck and trochanter from Baseline up to 6 months and 12 months | Baseline 、 Month 6 and Month 12
  Percent change in BMD at the total hip, femoral neck and trochanter as measured BMD is the amount of bone mineral in bone tissue. BMD scan was done using DXA. It is used to identify osteoporosis, determine risk for fractures, and measure response to osteoporosis treatment. The percentage change from Baseline for BMD was calculated as the value at the indicated time point minus the Baseline value multiplied by 100 and divided by the Baseline value.
Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) and Serum Procollagen Type I N Propeptideserum (s-PINP) from Baseline up to 6 months and 12 months | Baseline 、 Month 6 and Month 12
  s-CTX is biomarker of bone resorption and formation. s-CTX was assessed during Screening, Month 6 and Month 12 in the Double-blind Treatment Phase. The value during Screening was considered as the Baseline value. Percent change from Baseline was assessed as the value at the indicated visit minus the Baseline value divided by the Baseline value x 100.
  s-PINP is biomarker of bone resorption and formation. s-PINP was assessed during Screening, Month 6 and Month 12 in the Double-blind Treatment Phase. The value during Screening was considered as the Baseline value. Percent change from Baseline was assessed as the value at the indicated visit minus the Baseline value divided by the Baseline value x 100
Adverse events and serious adverse events | Baseline、 Month 1、 Month 3、 Month 6 、 Month 9 and Month 12
  Evaluation of the follwing parameters. Including adverse events(AEs), change in physical examination findings, change in vital signs, clinical laboratory testing for systemic safety,including liver function,renal function ,compelete blood count,and clinical chemistries
Immunogenicity | Baseline、 Month 3、 Month 6 、 Month 9 and Month 12
  Anti-denosumab antibody formation was assessed. Binding antibody and neutralizing antibody assays were used to assess number of participants with anti-denosumab antibody.

CONTACTS AND LOCATIONS:
Overall Officials: zhenlin zhang, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai sixth people's hospital, Shanghai, Shanghai Municipality, China